CLINICAL TRIAL: NCT04045431
Title: A Multi-centre Randomized, Controlled, Double-blind Clinical Investigation of Intra-articular Polyacrylamide Hydrogel in Subjects With Knee Osteoarthritis Followed by an Open Label Extension Study
Brief Title: Treatment of Knee Osteoarthritis With PAAG-OA
Acronym: ROSA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Contura (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CON-OA-001
Record Dates: First submitted 2019-07-08; First posted 2019-08-05 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2024-01

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: The subject and study staff will not know the treatment received. Only the unblinded injector will know the treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PAAG-OA (Experimental): Intra-articular injection with PAAG-OA (polyacrylamide hydrogel)
  Interventions: Device: PAAG-OA
- Synvisc-One (Active Comparator): Intra-articular injection with Synvisc-One (hyaluronic acid)
  Interventions: Device: Synvisc-One

INTERVENTIONS:
Device: PAAG-OA — Intra-articular injection of 6ml PAAG-OA in the target knee (incl. five (5) years follow-up) period.
  Arms: PAAG-OA
Device: Synvisc-One — Intra-articular injection of 6ml Synvisc-One in the target knee
  Arms: Synvisc-One

SUMMARY:
This is a multi-center, randomized, double-blind clinical investigation to compare the effectiveness of intra-articular polyacrylamide hydrogel (PAAG-OA) and a hyaluronic acid, Synvisc-One to induce symptomatic benefit in subjects with knee osteoarthritis.

DETAILED DESCRIPTION:
The trial is designed as a multi-center, randomised, controlled, double-blind, and parallel-group trial spanning over 12 months with outcome assessments at baseline, 1, 3, 6 and 12 months incl. follow-up period between 2-5 years. Primary endpoint at 6 months. The trial is designed to compare effectiveness and safety of injection of PAAG-OA and Synvisc-One® in participants with knee OA.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Male or female, aged ≥ 40 years
* Clinical diagnosis of knee OA American College of Rheumatology criteria confirmed by radiology
* Definite radiographic OA in the most symptomatic knee (target knee) at mild to moderate-stage (Kellgren-Lawrence grades 2 or 3)
* Stable dose of analgesics for the past four weeks
* NRS (11 points (0-10) pain intensity numerical rating scale) ≥ 4 in target knee, during the past week when walking
* Body Mass Index (BMI) between 20-35
* For females of reproductive potential: use of adequate contraception must be used throughout the trial

Exclusion Criteria:

* Female participants who are pregnant, lactating or planning pregnancy during the course of the clinical investigation
* Contraindications to PAAG-OA or Synvisc-One®, according to IB or Instruction for Use (IFU)
* Previous intra-articular injection of polyacrylamide gel in the target knee
* Previous intra-articular injection with hyaluronic acid or derivatives in target knee in the previous 6 months
* Significant valgus/varus deformity of the knee, ligamentous laxity or meniscal instability
* Other diseases in target knee than osteoarthritis
* Intra-articular injection of any substance other than hyaluronic acid (e.g. corticosteroids) in the target knee within the last 3 months
* Acute serious infection of any region that required hospital care or intravenous antibiotic treatment within the last 30 days, or oral antibiotic treatment within the last 14 days
* Skin disease or infections in the area of the injection site
* Infected or severely inflamed knees
* History of sepsis in any joint or any clinical concern for a subacute infectious process in the target knee
* History of surgery in the target knee within the past 6 months
* Symptomatic osteoarthritis of the hips, spine or ankle, that interferes with the evaluation of the target knee
* Planned surgery on any lower extremity
* Clinically significant venous or lymphatic stasis present in the legs
* Clinically apparent tense effusion or inflammation in the target knee
* Suffering from any unstable or severe cardio-vascular disease
* Any contraindication to intra-articular e.g. anticoagulant therapy or clinical concern for potential coagulopathy (e.g. liver disease)
* Any foreign material in the target joint
* Any significant medical condition (e.g. significant psychiatric or neurological disorders or active alcohol/drug abuse), any medical condition that is unstable/poorly controlled or other factors that may interfere with study participation
* Treatment with systemic steroids
* History of drug/alcohol abuse, mental dysfunction of other factors limiting their ability to cooperate fully
* Change in physiotherapy within the previous month
* Fibromyalgia
* Inflammatory or other disease/condition which may affect joints (e.g. rheumatoid arthritis, psoriatic arthritis and ankylosing spondylitis among others)
* Haemophilia
* Any other condition that in the opinion of the investigator put a potential participant at risk or otherwise precludes participation in the trial
* Known allergic reactions to components of Synvisc-One (avian protein)
* Known allergic reactions to antibiotics (azithromycin and moxifloxacin) or local anaesthesia
* Participation in any experimental device study within 6 months prior to enrolment, or participation in an experimental drug study within 1 month prior to enrolment

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 238 (Estimated)
Dates: Start 2019-05-15 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Comparing one injection of PAAG-OA with one injection of Synvisc-One on pain over 6 months in subjects with knee osteoarthritis | 6 months
  Change in WOMAC (WOMAC Osteoarthritis Index) pain subscale. Pain is reported in each of five response categories (0=none, 4=extreme)

SECONDARY OUTCOMES:
WOMAC | 1, 3, 6 and 12 months
  WOMAC (WOMAC Osteoarthritis Index) self reported pain, stiffness and physical function, categories (0=none, 4=extreme)
PGA (Patient Global Assessment) | 1, 3, 6 and 12 months
  PGA reported on a 10 cm Visual Analogue Scale
EQ-5D-5L, QoL | 1, 3, 6 and 12 months
  EQ-5D-5L, Quality of Life, comprised of descriptive system where each dimension has 5 levels (ranging from no problems to extreme problems) and a 20 cm Visual Analogue Scale (0 = worst health and 100 = best health)
OMERACT-OARSI responder criteria | 1, 3, 6 and 12 months
  Per the OMERACT-OARSI criteria, a subject is classified as a positive responder if at least one (1) of the following two (2) conditions is observed at the post-baseline assessment:
  * In either pain (WOMAC pain subscale) or function (WOMAC function subscale), a high improvement in the subscale, where high improvement in a subscale is achieved if there is both a > 50% improvement from Baseline and an absolute change from Baseline of > 20 normalised units (0-100 scale) OR
  * Improvement in at least two (2) of the following three (3):
    1. Improvement in pain (WOMAC pain subscale) defined as > 20% improvement from Baseline and an absolute change from Baseline of > 10 (0-100 scale)
    2. Improvement in function (WOMAC function subscale) defined as > 20% improvement from Baseline and an absolute change from Baseline of > 10 (0-100 scale)
    3. Improvement in PGA defined as > 20% improvement from Baseline and an absolute change from Baseline of > 10 mm (0-100 sc

CONTACTS AND LOCATIONS:
Overall Officials: Henning Bliddal, MD, Principal Investigator — The Parker Institute
Locations (3):
- Denmark (3):
  - The Parker Institute, Frederiksberg
  - A2 Reumatologi og idrætsmedicin, Hillerød
  - Reumatolog i Odense, Odense

REFERENCES:
- [Derived] Bliddal H, Beier J, Hartkopp A, Conaghan PG, Henriksen M. Three-year follow-up from a randomised controlled trial of a single intra-articular polyacrylamide hydrogel injection in subjects with knee osteoarthritis. Clin Exp Rheumatol. 2025 Dec 11. doi: 10.55563/clinexprheumatol/5lofry. Online ahead of print. PMID 41487107